CLINICAL TRIAL: NCT01953666
Title: Phase 1 Evaluation of the Influence of Settings of Word Prediction Software (Phase 1)and the Efficiency of Rehabilitation Programm (Phase 2)to Text Input Speed for People With Spinal Cord Injury
Brief Title: Evaluation of the Efficiency of Word Prediction Software to Text Input Speed for Tetraplegia
Acronym: Smartwrite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Pouplin Samuel, ergotherapeute (Occupational Therapist), Centre d'Investigation Clinique et Technologique 805
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12053
Record Dates: First submitted 2013-09-17; First posted 2013-10-01 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Settings Word Prediction Software; Rehabilitation Program
Keywords: word prediction software, text input speed, copm, occupational therapist, rehabilitation, spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rehabilitation Group (Experimental): People with spinal cord injury who have a rehabilitation program on a word prediction software with an occupational therapist.
  Interventions: Other: Rehabilitation program
- Self Training at Home Group (Active Comparator): People with spinal cord injury who don't have a rehabilitation program with an occupational therapist but who have instructions for learning at home on a word prediction software
  Interventions: Other: Self - Training at home
- No treatment Group (No Intervention): People with spinal cord injury who don't have instructions, rehabilitation programm on word prediction software. They have no treatment.

INTERVENTIONS:
Other: Rehabilitation program — Rehabilitation program with an occupational therpasit
  3 training sessions (one hour) per week for a month (12 sessions)
  Arms: Rehabilitation Group
Other: Self - Training at home — Only instructions for a self - training at home
  Arms: Self Training at Home Group

SUMMARY:
Computers now play an important role in the lives of most individuals.Access to computers is crucial for people with disabilities and may improve their quality of life. The use of computers can facilitate mainstreaming at school, for example, and the Internet may provide a valuable means of communication. However, the use of computers requires a certain degree of motor ability. People with motor disabilities frequently experience difficulties using a standard keyboard and standard pointing input systems such as a mouse. Many solutions exist to facilitate computer access, depending on the person's specific impairments and the purpose for which the computer is used. The most common solution relies on the use of a virtual keyboard which is directly displayed on the computer screen. The selection of the desired key on the virtual keyboard can be handled by a large variety of input devices, from a microgravity mouse to single switch devices supplemented by a process of dynamic scanning of the keyboard.Although such assistive devices render computers accessible to people with disabilities, the actual inputting of text can be very slow. A method to increase text input speed is to display words which are predicted from the letters previously typed. Word prediction reduces the number of necessary key strokes by avoiding having to type the whole word. The effect on text input speed is, however uncertain and results in the literature are inconclusive. Indeed, word prediction software provide a enhancement of cognitive load which decrease text input speed.The reduction of cognitive load could therefore be based in part on the optimization settings of the software and / or achievement of a rehabilitation program.Our hypothesis are for people with spinal cord injury : i) optimization settings word prediction software and ii) a rehabilitation program could improve the text input speed.The investigators propose to study the influence of settings word prediction software on text input speed and the influence of a rehabilitation program provided by a therapist, focused on word prediction software to help integrate them. The aim is to increase the performance of people with spinal cord injury and their satisfaction.

The first phase of this research is to select the word prediction software and configuration that provides the best user support.The second phase corresponds to the objective of evaluating the efficiency of a rehabilitation program .

DETAILED DESCRIPTION:
PHASE 1 : The first phase studied the repeated measurement of the efficiency of typing text topics in various situations. Each subject will copy a text different in each test and in a random order. Similarly, if the word prediction software has a capacity for self-improvement the internal dictionary, it will be disabled.

the investigators will study one setting of the configuration word prediction software. Are available the length of the list of proposals for which three options are selected: 1, 3 or 5 words, according to the literature and to the results of a questionnaire.This questionnaire was sent to identify the use of people with spinal cord injury and professionals about word prediction software.

The list of words is in the upper position of the screen based on the results of the questionnaire.

Four combinations will be tested on each subject. Twelve Tetraplegics will be required in each group (one group using a virtual keyboard and one group using the physical keyboard) Each combination will be tried for 10 minutes.

PHASE 2 :

The second phase will evaluate the effeciency of a rehabilitation program reduced cognitive load generated by the software predictions words.

The investigators propose an evaluation of the effects of 12 training sessions in a controlled, randomized, three parallel groups (experimental group : rehabilitation program, a group : a self-learning and a group : no learning).

Text input tests will be performed before and after the training sessions for people who have rehabilitation program. For the other two groups, those will be reviewed one month after the first test.

For this evaluation, a different text but with the same difficulty will be used. The order of execution will be randomized.

At the end of the month the three groups will be evaluated according to the same procedures for the firts test.

ELIGIBILITY:
Inclusion Criteria:

* Tetraplegia (between C4 and C8 ASIA) more than 6 months.
* Can read and write
* No visual problems preventing the use of computers.
* Recipient of a Health Insurance Plan
* Having read information note.

Exclusion Criteria:

* Moving in progress or predictable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from Text Input Speed at 1 month | Phase 1 After every test (10 minutes) Phase 2 : 1 months
  text input speed (characters/minute)

SECONDARY OUTCOMES:
Change from Errors at 1 month | Phase 1 After every test (10 minutes) Phase 2 : 1 month
  We record errors in text entry test
Change from Prediction use at 1 month | Phase after every test (10 minutes) Phase 2 : 1 month
  Number of use of word prediction software
Change from Satisfaction | Phase 1 After every test (10 minutes) Phase 2 : 1 month
  Satisfaction of people with spinal cord injury about word prediction software (visual analogue scale)
Change from Cognitive load at 1 month | Phase 1 After every test (10 minutes) Phase 2 : 1 month
  Cognitive load of people with spinal cord injury (visual analogue scale)
Change from Speed sensation at 1 month | Phase 1 After every test (10 minutes) Phase 2 : 1 month
  speed sensation of people with spinal cord injury with word prediction software (visual analogue scale)

CONTACTS AND LOCATIONS:
Overall Officials: Djamel Bensmail, MDPHD, Study Director — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, France